CLINICAL TRIAL: NCT00312221
Title: Randomized, Double-blind, Multicenter Study to Determine the Efficacy and Safety of BTDS 20 or Oxycodone Immediate-Release (OxyIR) Versus BTDS 5 in Subjects With Moderate to Severe Osteoarthritis (OA) Pain
Brief Title: Safety and Efficacy of Buprenorphine Transdermal System (BTDS) in Subjects With Moderate to Severe Osteoarthritis Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated early for administrative reasons unrelated to safety or efficacy
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUP3019
Record Dates: First submitted 2006-04-06; First posted 2006-04-07 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, opioid, transdermal
MeSH Terms: conditions — Osteoarthritis | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BTDS 5 (Active Comparator): Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
  Interventions: Drug: Buprenorphine
- BTDS 20 (Experimental): Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
  Interventions: Drug: Buprenorphine
- Oxycodone Immediate-Release (Oxy IR) 40 mg (Experimental): Oxycodone immediate-release 40 mg (two 5-mg capsules every 6 hours).
  Interventions: Drug: oxycodone immediate-release

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
  Other Names: Butrans™
  Arms: BTDS 5
Drug: Buprenorphine — Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
  Other Names: Butrans™
  Arms: BTDS 20
Drug: oxycodone immediate-release — Oxycodone immediate-release 40 mg (two 5-mg capsules every 6 hours).
  Arms: Oxycodone Immediate-Release (Oxy IR) 40 mg

SUMMARY:
The objective of this study is to demonstrate the effectiveness and tolerability of the buprenorphine transdermal system (20 mg) in comparison to the buprenorphine transdermal system (5 mg) and oxycodone immediate release in subjects with moderate to severe osteoarthritis pain currently treated with oral opioids. The double-blind treatment intervention duration is 12 weeks during which time supplemental analgesic medication (acetaminophen, ibuprofen, immediate release oxycodone) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the hip, knee, or spine for 1 year or longer, confirmed by radiographic evidence within the last 2 years.
* Good pain control while on a stable dose of an opioid analgesic for osteoarthritis.

Exclusion Criteria:

* Not currently taking and tolerating opioids.
* Taking more than 80 mg per day of oral morphine sulfate or equivalent within 30 days of enrollment.
* Requiring frequent analgesic therapy for chronic condition(s), in addition to osteoarthritis.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2004-04; Primary Completion 2005-07 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Parkway Medical Center, Birmingham, Alabama
  - International Clinical Research Network, Chula Vista, California
  - Clinical Trials Research, Roseville, California
  - Accelovance, San Diego, California
  - Torrance Clinical Research, Torrance, California
  - Southern Colorado Clinic, Pueblo, Colorado
  - Drug Study Institute, Jupiter, Florida
  - Innovative Research of West Florida, Inc., Largo, Florida
  - International Medical Research, Ormond Beach, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Georgia Medical Research Institute, Marietta, Georgia
  - Non- Surgical Orthopedic & Spine Center, P.C., Marietta, Georgia
  - The Arthritis Center, Springfield, Illinois
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Miray Medical Center, Brockton, Massachusetts
  - Professional Clinical Research Crystal Lake Health Center, Benzonia, Michigan
  - Rheumatology PC, Kalamazoo, Michigan
  - Pharm Quest, Greensboro, North Carolina
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Med Search Professional Group/Pharmaceutical C-Trials Inc., Hurst, Texas
  - Texas Medical Research Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Dates: 02-Apr-2004 (first subject first visit) to 18 Jul-2005 (last subject last visit); 15-Jun-2005 (first site notified of study termination). The study took place in 82 medical/research sites in the US; 59 sites randomized at least 1 subject.
Pre-assignment Details: Men and women aged 40 years or older with OA of the hip, knee, or spine, on 30 to 80 mg/day morphine sulfate (MSO4) or equivalent, with or without nonopioid analgesic medication. (652 subjects entered the run-in period; 418 completed.) Subjects were eligible to enter the double-blind phase if they tolerated BTDS 20 and achieved stable analgesia.
Groups:
- Run-in Period: The run-in period was designed to select subjects whose pain was adequately controlled by and who tolerated BTDS 20 treatment. BTDS 10 or 20 was applied for 7-day wear during the 3-week run-in period.
- Double-blind BTDS 5: Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
- Double-blind BTDS 20: Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
- Double-blind Oxycodone Immediate-Release: Oxycodone immediate-release 40 mg (two 5-mg capsules every 6 hours).
Period: Open-label Run-in Period
Arm/Group | Run-in Period | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Started | 652 | 0 | 0 | 0
Completed | 418 | 0 | 0 | 0
Not Completed | 234 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0
Not completed — Adverse Event | 74 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 0
Not completed — Administrative | 42 | 0 | 0 | 0
Not completed — Lack of Efficacy | 102 | 0 | 0 | 0
Not completed — Did not qualify | 5 | 0 | 0 | 0
Period: Double-blind Phase
Arm/Group | Run-in Period | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Started | 0 | 136 | 149 | 133
Completed | 0 | 77 | 77 | 63
Not Completed | 0 | 59 | 72 | 70
Not completed — Withdrawal by Subject | 0 | 6 | 8 | 7
Not completed — Adverse Event | 0 | 10 | 19 | 18
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Administrative | 0 | 26 | 37 | 33
Not completed — Lack of Efficacy | 0 | 17 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release | Total
Number analyzed (Participants) | 136 | 149 | 133 | 418
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.71) | 57.9 (9.45) | 58.1 (10.36) | 58.3 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 116 | 94 | 311
  Male | 35 | 33 | 39 | 107

OUTCOME MEASURES:

1. Primary Outcome: "Average Pain Over the Last 24 Hours" Scores at Weeks 4, 8, and 12 of the Double-blind Phase.
Description: The "average pain over the last 24 hours" score was collected using an 11-point numerical scale ranging from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. This variable was obtained at each clinic visit during the double-blind phase of the study (postrandomization weeks 1, 2, 4, 8, and 12).
Time Frame: Weeks 4, 8, and 12 of the double-blind phase
Population: Full Analysis Population (N = 418) consisted of subjects who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 136 | 149 | 133
Units on a scale
  Screening | 6.60 (0.116) | 6.58 (0.103) | 6.44 (0.117)
  Prerandomization | 3.25 (0.114) | 3.02 (0.093) | 3.03 (0.099)
  Week 4 | 4.21 (0.219) | 3.57 (0.195) | 3.45 (0.209)
  Week 8 | 3.78 (0.239) | 3.37 (0.190) | 3.59 (0.217)
  Week 12 | 3.67 (0.246) | 3.56 (0.230) | 3.37 (0.232)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.8562 to 0.1054] — Treatment comparison between BTDS 20 and BTDS 5 during the 12-week double-blind phase
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; Test type: Superiority or Other; p = 0.140, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI [-0.8455 to 0.1189] — Treatment comparison between BTDS 5 and oxycodone immediate-release during the 12-week double-blind phase

2. Secondary Outcome: The Mean Daily Number of Supplemental Analgesic Medication Tablets
Description: The mean daily number of supplemental analgesic medication tablets included sponsor-supplied ibuprofen, acetaminophen, or OxyIR®.
Time Frame: Double-blind phase (84 days)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Tablets
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 136 | 149 | 133
Tablets
  Prerandomization | 2.0 (0.19) | 1.7 (0.13) | 1.6 (0.13)
  Double-blind | 3.3 (0.26) | 2.3 (0.19) | 2.3 (0.22)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.47 to -0.20] — Treatment comparison between BTDS 5 and BTDS 20 during the 12-week double-blind phase
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; Test type: Superiority or Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.47 to -0.17] — Treatment comparison between BTDS 5 and oxycodone immediate-release during the 12-week double-blind phase

3. Secondary Outcome: The Physical Function Subscale of The Western Ontario and McMaster's Universities Osteoarthritis (WOMAC OA) Index at Weeks 4, 8, and 12 of the Double Blind Phase
Description: The WOMAC (Version LK 3.1) measures symptoms and physical functioning of patients with OA of the hip and knee. It contains 24 items (5 pain, 2 stiffness, 17 physical function) and takes less than 5 minutes to complete.
  The WOMAC physical function subscale has 17 items coded as 0 to 4 (best to worst), which are summed, giving a range of 0 to 68 (best to worst).
Time Frame: Weeks 4, 8 and 12 of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 136 | 149 | 133
Units on a scale
  Screening | 36.88 (1.093) | 37.69 (0.930) | 36.81 (1.043)
  Prerandomization | 25.96 (0.993) | 24.19 (0.947) | 24.42 (0.930)
  Week 4 | 30.60 (1.187) | 28.34 (1.025) | 26.65 (1.253)
  Week 8 | 28.70 (1.364) | 28.34 (1.199) | 26.59 (1.405)
  Week 12 | 29.68 (1.500) | 29.35 (1.253) | 27.25 (1.651)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; Test type: Superiority or Other; p = 0.707, Mixed Models Analysis; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-3.0054 to 2.0397] — Treatment comparison between BTDS 5 and BTDS 20 during the 12-week double-blind phase
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; Test type: Superiority or Other; p = 0.187, Mixed Models Analysis; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-4.4459 to 0.8706] — Treatment comparison between BTDS 5 and oxycodone immediate-release during the 12-week double-blind phase

4. Secondary Outcome: The Sleep Disturbance Subscale in The Medical Outcomes (MOS)-Sleep Scale at Weeks 4, 8, and 12 of the Double-blind Phase
Description: The MOS-Sleep Scale consists of 12 individual items: (4 sleep disturbance, 2 sleep adequacy, 1 quantity of optimal sleep, 3 somnolence, 1 snoring, and 1 shortness of breath) and takes 5 to 10 minutes to complete. Question 1 is scored on a scale of 1 to 5 and Questions 2 to 12 are scored on a scale of 1 to 6. The Sleep Disturbance Subscale score is derived from the scores to Questions 1, 3, 7 and 8, and ranges from 0 to 100, where higher scores indicate greater sleep disturbance.
Time Frame: Weeks 4, 8, and 12 of the Double-blind Phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 136 | 149 | 133
Units on a scale
  Screening | 51.91 (2.139) | 55.28 (2.035) | 55.74 (2.197)
  Prerandomization | 34.64 (1.950) | 28.65 (1.782) | 33.03 (1.926)
  Week 4 | 39.23 (2.144) | 32.40 (1.941) | 35.72 (2.298)
  Week 8 | 35.95 (2.791) | 31.71 (2.473) | 34.13 (2.746)
  Week 12 | 39.13 (3.089) | 32.95 (2.819) | 36.32 (3.290)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; Test type: Superiority or Other; p = 0.685, Mixed Models Analysis; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-5.6177 to 3.6930] — Treatment comparison between BTDS 5 and BTDS 20 during the 12-week double-blind phase
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; Test type: Superiority or Other; p = 0.443, Mixed Models Analysis; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-6.4415 to 2.8255] — Treatment comparison between BTDS 5 and oxycodone immediate-release during the 12-week double-blind phase

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) occurring after the signing of informed consent up to study completion or discontinuation; during 7 days after last visit; serious AEs up to 30 days following the last study visit were followed until the event resolved.
Description: AEs were obtained through spontaneous reports and subject interview.
Groups:
- Double-blind BTDS 5: Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear during the 12-week double-blind phase
- Double-blind BTDS 20: Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear during the 12-week double-blind phase
- Double-blind Oxycodone Immediate-Release: Oxycodone immediate-release 40 mg (two 5-mg capsules every 6 hours) during the 12-week double-blind phase.
- Run-in, Open-label BTDS 10 and 20: The run-in period was designed to select subjects whose pain was adequately controlled by and who tolerated BTDS 20 treatment. BTDS 10 or 20 was applied for 7-day wear during the 3-week run-in period.
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release | Run-in, Open-label BTDS 10 and 20
Serious Adverse Events (participants affected / at risk) | 3/136 | 7/149 | 7/133 | 8/652
Other Adverse Events (participants affected / at risk) | 30/136 | 70/149 | 56/133 | 187/652
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind BTDS 5 (N=136) | Double-blind BTDS 20 (N=149) | Double-blind Oxycodone Immediate-Release (N=133) | Run-in, Open-label BTDS 10 and 20 (N=652)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Chest pain with ischemic episode (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Dermoid ovarian cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Enlarged uterus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Exacerbation of Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Exacerbation of lumbar spinal stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment "Fall" and "Fell" are listed as 2 separate categories.
Fell (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment "Fall" and "Fell" are listed as 2 separate categories.
Fractured left hip (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
GI bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Muscle spasms right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
OxyIR abuse (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessment
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments.
Paroxysmal supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments.
Postsurgical hip joint dislocation, left hip (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Possible bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments.
Prostatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Recurrent L4-L5 disc herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments.
Recurrent L5-S1 disc herniation with impingement of the S1 nerve root (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments.
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments.
Transischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments.
Worsening asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments.
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments.
End stage OA of the right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind BTDS 5 (N=136) | Double-blind BTDS 20 (N=149) | Double-blind Oxycodone Immediate-Release (N=133) | Run-in, Open-label BTDS 10 and 20 (N=652)
Nausea (Gastrointestinal disorders) | 4 | 16 | 17 | 94 — Systematic and nonsystematic assessments
Constipation (Gastrointestinal disorders) | 3 | 8 | 9 | 22 — Systematic and nonsystematic assessments
Vomiting NOS (Gastrointestinal disorders) | 0 | 8 | 6 | 32 — Systematic and nonsystematic assessments
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 6 | 1 — Systematic and nonsystematic assessments
Application site pruritus (General disorders) | 13 | 22 | 12 | 47 — Systematic and nonsystematic assessments
Application site rash (General disorders) | 5 | 9 | 8 | 9 — Systematic and nonsystematic assessments
Application site erythema (General disorders) | 9 | 14 | 5 | 9 — Systematic and nonsystematic assessments
Pain NOS (General disorders) | 5 | 1 | 7 | 11 — Systematic and nonsystematic assessments.
Upper respiratory tract infection NOS (Infections and infestations) | 6 | 6 | 8 | 5 — Systematic and nonsystematic assessments.
Urinary tract infection NOS (Infections and infestations) | 5 | 8 | 5 | 9 — Systematic and nonsystematic assessments.
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 4 | 12 — Systematic and nonsystematic assessments.
Pain in limb (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3 | 14 — Systematic and nonsystematic assessments.
Headache (Nervous system disorders) | 10 | 22 | 16 | 70 — Systematic and nonsystematic assessments.
Dizziness (Nervous system disorders) | 4 | 10 | 7 | 43 — Systematic and nonsystematic assessments.
Somnolence (Nervous system disorders) | 2 | 2 | 10 | 29 — Systematic and nonsystematic assessments.

LIMITATIONS AND CAVEATS:
This study was terminated early for administrative reasons not related to safety or efficacy. Low enrollment at termination led to reduced power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days